CLINICAL TRIAL: NCT04214925
Title: Investigation of the Effectiveness of Tai Chi Exercise Program on Trunk Endurance, Balance, Sleep, Fatigue, Anxiety and Depression in Scleroderma Patients: A Randomized Controlled Study
Brief Title: Effectiveness of Tai Chi Exercise Program in Scleroderma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Bilge Basakci Calik, Assoc Prof, PT, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60116787-020 / 20653
Record Dates: First submitted 2019-12-25; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Tai Chi
Keywords: Scleroderma; Tai Chi; sleep; fatique; depression; anxiety
MeSH Terms: conditions — Scleroderma, Diffuse; Depression; Anxiety Disorders | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: randomized controlled parallel group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of Tai Chi intervention (Experimental): Tai Chi exercise program will create by selecting the first-basic 10 forms from 24 short forms of Yang style. The forms' name: Beginning, Parting the Horse's Mane, Stork Spreading Its Wings, Brushing Your Knees and Stepping, Playing The Pipes, Fending Off the Monkey, Grasping the Sparrow's Tail Left, Grasping the Sparrow's Tail Right, Simple Whip, Moving Hands Like Clouds-Conclusion. All forms will be completed at 10 weeks. Each session will take 1 hour (15 min for warming up exercises, 30 min of Tai Chi forms, and 15 min for cooling down exercises). The 14 patients of SS in this group will be divided into two groups of 7.
  Interventions: Other: Tai Chi
- Group of home exercises (Other): The home exercise group will receive a one-hour home program, 2 days a week. The first and last 15 minutes of the exercise program will consist of warm-up and cooling- down exercises. After warm-up exercises, stretching for shoulder, hamstring and erector spinae muscles, strengthening exercises for abdominal and back muscles will be performed 10 times each for 30 minutes.
  Interventions: Other: Tai Chi

INTERVENTIONS:
Other: Tai Chi — Home exercises will include warm-up and cool-down exercises, stretching for shoulder, hamstring and erector spinae muscles, strengthening exercises for abdominal and back muscles.
  Other Names: Home exercises

SUMMARY:
Because of multiple system involvement, patients with Scleroderma have complaints such as fatigue, sleep disturbances, functional limitations, skin deformations, pain, swollen hands and joint pain. The aim of this study is to investigate the effect of Tai Chi exercise program on trunk endurance, balance, sleep, fatigue, anxiety and depression in patients with scleroderma.

DETAILED DESCRIPTION:
In the study, which will be planned as a randomized controlled parallel group, the effects of Tai Chi in SS patients are compared with the home exercise group. Evaluations before and after the treatment will make by a physiotherapist. Training of Tai Chi will supervised by an experienced and certified physiotherapist.

Lateral Bridge Test , Berg Balance Scale, Pittsburg Sleep Quality Index , Fatigue Severity Scale and Fatigue Impact Scale , Hospital Anxiety and Depression Scale will be used evaluation before and after training.

ELIGIBILITY:
Inclusion Criteria:

* have been diagnosed with scleroderma,
* have been sedentary (have not routinely participated in exercise activities during the past 3 months)
* have been using a fixed dose of medication for at least 6 months
* no communication problems
* having stable disease

Exclusion Criteria:

* a diagnosis of pulmonary hypertension
* a history of active infection, cardiac involvement, psychiatric disorder, a history of active myositis, renal failure, metastatic cancer, pregnancy
* Data of the participant whose changes were made during the study are not included in this study and participation is terminated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index | ten weeks
  The scale has 19 items and measures 7 components of sleep quality: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction (each domain score ranges between 0 and 3). A global PSQI score corresponding to the total of the individual scores from the 7 components is calculated (range = 0-21). A result equal to 6 or above is considered indicative of poor sleep quality. The test has high diagnostic specificity for detecting clinical sleep impairment.
Fatigue Severity Scale | ten weeks
  Fatigue Severity Scale comprises nine statements, describing the severity and impact of fatigue, with a scale of possible responses ranging from 1 ("strongly disagree") to 7 ("strongly agree"). FSS total scores are usually reported as the mean score over the nine items; a higher score indicates greater severity.
Fatigue Impact Scale | ten weeks
  It is a scale that evaluates the effects of fatigue on daily life activities and quality of life. It contains 40 questions in total. Consists of cognitive, physical and social subdivisions. The score ranges from 0 to 160 points and the high score indicates a negative impact.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | ten weeks
  It is a scale that evaluates the anxiety and depression levels of individuals in 14 questions. While the answers score between 0 and 3, the high score indicates high anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ayan, Dr, Study Director — Antalya Training and Research Hospital
Locations (1):
- Pamukkale University, Denizli, Kinikli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data are analyzed with SPSS (22.0 version) package program. Descriptive statistics will be presented as mean ± standard deviation (SD), number (n), and percentage (%).

REFERENCES:
- [Background] Mitropoulos A, Gumber A, Crank H, Akil M, Klonizakis M. The effects of upper and lower limb exercise on the microvascular reactivity in limited cutaneous systemic sclerosis patients. Arthritis Res Ther. 2018 Jun 5;20(1):112. doi: 10.1186/s13075-018-1605-0. PMID 29871697